CLINICAL TRIAL: NCT02351154
Title: Grading Atrophic Gastritis by a New Quantitative Method Using Confocal Laser Endomicroscopy Probe (p-CLE): First Results of a Prospective Cohort Study
Brief Title: Grading Atrophic Gastritis by Confocal Laser Endomicroscopy Probe (p-CLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IECED 01-08-2014
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atrophic gastritis (Other): gastric glands (crypts) with atrophic gastritis were measured using the Cellvizio Viewer software
  Interventions: Other: Cellvizio Viewer software

INTERVENTIONS:
Other: Cellvizio Viewer software — permets to perform analysis of diameters in micrometers

SUMMARY:
Atrophic gastritis (AG) is a chronic disease, associated to gastric adenocarcinoma moreover if severity AG is present. Sydney system classified AG as mild, moderate and severe, but with moderate interobserver agreement, due to this system is based in a visual analogic scale (qualitative analysis). Confocal endomicroscopy showed an accuracy of 98% for diagnosis gastric diseases, but when grading AG still remains a qualitative measure. Recently, a new software called "Cellvizio® Viewer" (CV) permits to measure in micrometers (µm) the structures observed after confocal laser endomicroscopy probe studies. Based on the hypothesis that AG severity is correlated with crypts size diminution, the aim of this study is to determine a quantitative way to classify the severity of AG measuring the crypt area and inter-crypt spaces in patients with AG.

DETAILED DESCRIPTION:
Consecutive patients that underwent to upper endoscopy (UE) evaluation were included in this study. All subjects went to UE according to standard procedure, under propofol sedation, and using a high definition endoscope with a working channel of 2.8 mm After gastric mucosa inspection using endoscopy, in vivo microscopy analysis at x1000 magnification was done using confocal laser endomicroscopy probe (p-CLE) in all patients.

During UE 5 biopsy sites were performed in accordance to update Sydney system first using p-CLE and them by biopsy forceps from the same site (2 from the lesser and greater curvature of the antrum about 2-3 cm near the pylorus, 2 from the middle portion of the lesser and greater curvatures of the corpus about 8 cm from the cardia, and 1 from the angulus). p-CLE images were recorded as video frames and pictures during in vivo microscopy analysis.

For histopathology all specimens were fixed in 10% formalin. An experienced histopathologist analyzed the histological features of each sample with hematoxylin and eosin staining and made the diagnosis according to the updated Sydney classification.

At p-CLE normal crypt was defined by using the classification of Wang et al. After histopathology confirm GA, crypts were analyzed using the CV software that is a post-procedure tool that could be installed in computers, working as a laboratory data analyzer. This software permits to measure diameters of the microscopy findings in an escalade model in micrometers, using different colors lines and giving their results in a table that could be exported as excel table for analysis of the results The crypts diameters were measuring to determine the area by using the elliptic area formula (A = π.d1.d2). The inter-crypt space was also measured and defined as the mean of each measured distance between the studied crypt and it's adjacent.

The cutoff value between mild, moderate and severe GA, crypts area was classified across tertiles, expressing its distribution using a box-spot graphic. For relationship between crypt area (CA) and inter-crypt space, quadratic polynomial regression was used. Data was processed using IBM® SPSS® Statistics.

ELIGIBILITY:
Inclusion Criteria:

* dyspepsia >12 months
* age ≥18, no history of UE evaluation
* GA at histopathology
* acceptance to participate.

Exclusion Criteria:

* use of proton pump inhibitors
* antibiotics or NSAID´s
* gastric cancer
* gastric surgery
* pregnancy
* contraindication to fluorescein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Gastric crypt diameters | 3 months
  to determine the area of the gastric crypt measured by the elliptic area formula (A = π.d1.d2)

SECONDARY OUTCOMES:
Gastric inter-crypt diameters | 3 months
  measuring the distance of the gastric inter-crypt space.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Result] Wang P, Ji R, Yu T, Zuo XL, Zhou CJ, Li CQ, Li Z, Li YQ. Classification of histological severity of Helicobacter pylori-associated gastritis by confocal laser endomicroscopy. World J Gastroenterol. 2010 Nov 7;16(41):5203-10. doi: 10.3748/wjg.v16.i41.5203. PMID 21049554
- [Result] Zhang JN, Li YQ, Zhao YA, Yu T, Zhang JP, Guo YT, Liu H. Classification of gastric pit patterns by confocal endomicroscopy. Gastrointest Endosc. 2008 May;67(6):843-53. doi: 10.1016/j.gie.2008.01.036. PMID 18440377
- [Result] Dixon MF, Genta RM, Yardley JH, Correa P. Classification and grading of gastritis. The updated Sydney System. International Workshop on the Histopathology of Gastritis, Houston 1994. Am J Surg Pathol. 1996 Oct;20(10):1161-81. doi: 10.1097/00000478-199610000-00001. PMID 8827022